CLINICAL TRIAL: NCT01453439
Title: CBT Versus Supportive Psychotherapy for Body Dysmorphic Disorder
Brief Title: Cognitive-Behavioral Therapy and Supportive Psychotherapy for Body Dysmorphic Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Sabine Wilhelm, PhD, Sabine Wilhelm, PhD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH091078 (NIH); R01MH091078 (NIH); 2010-P-001021/2 (Other: Institutional Review Board)
Record Dates: First submitted 2011-08-30; First posted 2011-10-17 (Estimated); Results first posted 2020-07-15 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Body Dysmorphic Disorder; Obsessive-Compulsive Spectrum Disorder; Anxiety Disorders; Somatoform Disorders
Keywords: Body dysmorphic disorder; Obsessive compulsive spectrum disorder; Body image; Appearance concerns
MeSH Terms: conditions — Body Dysmorphic Disorders; Anxiety Disorders; Somatoform Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Behavioral Therapy (Experimental): Group receiving Cognitive-Behavioral Therapy
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Supportive Psychotherapy (Active Comparator): Group receiving Supportive Psychotherapy
  Interventions: Behavioral: Supportive Psychotherapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Participants will receive a total of 22 sessions (over 24 weeks) of individual, manual-based CBT. During the sessions, participants will receive education about BDD and CBT, learn to develop more helpful thoughts and beliefs, gradually enter anxiety provoking situations while reducing compulsions (repetitive behaviors), and learn relapse prevention techniques.
  Other Names: CBT
  Arms: Cognitive Behavioral Therapy
Behavioral: Supportive Psychotherapy — Participants will receive a total of 22 sessions (over 24 weeks) of individual, manual-based SPT. During the sessions, participants will receive education about BDD and SPT, learn about factors that may affect their symptoms (for example, relationships, work, stress), and learn to cope with challenges in their life by improving self-esteem and positive coping skills.
  Other Names: SPT
  Arms: Supportive Psychotherapy

SUMMARY:
The purpose of this study is to learn more about two different types of psychotherapy to help individuals who have body dysmorphic disorder (BDD). BDD is a severe, often chronic, and common disorder consisting of distressing or impairing preoccupation with perceived defects in one's physical appearance. Individuals with BDD have very poor psychosocial functioning and high rates of hospitalization and suicidality. Because BDD differs in important ways from other disorders, psychotherapies for other disorders are not adequate for BDD. Despite BDD's severity, there is no adequately tested psychosocial treatment (psychotherapy) of any type for this disorder. This study will compare the effectiveness of Cognitive Behavioral Therapy and Supportive Psychotherapy as well as predictors of improvement.

DETAILED DESCRIPTION:
Body Dysmorphic Disorder (BDD) is a common and severe disorder in which a person is preoccupied by perceived defects in his or her appearance. The purpose of this research study is to learn more about two different forms of therapy to help individuals with BDD: cognitive behavioral therapy (CBT), a promising new treatment for BDD, and supportive psychotherapy (SPT), the most commonly received therapy for BDD. The investigators would like to find out which treatment is more effective for BDD. The investigators will also examine patient characteristics that may predict response to treatment.

Participants will be randomly assigned (like the flip of a coin) to receive 22 sessions (over 24 weeks) of either CBT or SPT. Both treatments teach participants about BDD. CBT focuses on helping participants to develop more adaptive thoughts and beliefs and to gradually reduce avoidance and compulsive (repetitive) behaviors. SPT focuses on relationships, feelings, and other factors that may affect BDD symptoms (e.g., work, stress), and helps participants to cope with challenges in their life by improving self-esteem and positive coping.

For each participant, this study will last for 12 months. CBT and SPT sessions occur for 22 sessions over 24 weeks. The severity of participants' BDD-related symptoms and other symptoms will be assessed at the end of treatment (week 24), and at 3- and 6-months after treatment ends.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient men and women age 18 and older
* DSM-IV BDD or its delusional variant for at least 6 months
* BDD is the most problematic psychiatric disorder (in the patient's and clinician's opinion) and the primary reason for seeking treatment
* Score of 24 or higher on the BDD-Yale-Brown Obsessive Compulsive Scale

Exclusion Criteria:

* Current clinically significant suicidality and/or score on the BDI-II suicide item (#9) > 1
* Any clinical features requiring a higher level of care
* Mental retardation or borderline intellectual functioning (estimated IQ < 80 on the Wechsler Abbreviated Scale of Intelligence) or dementia, brain damage, or other cognitive impairment that would interfere with ability to engage in CBT
* DSM-IV substance abuse or dependence within the past 3 months; or a positive urine drug screen for any illicit substances of abuse
* Current manic episode
* Psychotic disorder
* Borderline personality disorder
* Body image concerns accounted for by an eating disorder
* Previous treatment with > 10 sessions of CBT for BDD
* Subjects cannot be receiving any other psychotherapy or begin such treatment during the study
* Patients can be receiving psychotropic medication if they have taken a stable dose for at least two months before the study baseline assessment and the dose remains stable during the study.
* Presence of any behavior (e.g., violence) that would interfere with full cooperation with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-08; Primary Completion 2017-01-05 (Actual); Study Completion 2017-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Wilhelm, Ph.D., Principal Investigator — Massachusetts General Hospital; Katharine Phillips, M.D., Principal Investigator — Rhode Island Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Rhode Island Hospital, Providence, Rhode Island

REFERENCES:
- [Derived] Wilhelm S, Phillips KA, Greenberg JL, O'Keefe SM, Hoeppner SS, Keshaviah A, Sarvode-Mothi S, Schoenfeld DA. Efficacy and Posttreatment Effects of Therapist-Delivered Cognitive Behavioral Therapy vs Supportive Psychotherapy for Adults With Body Dysmorphic Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2019 Apr 1;76(4):363-373. doi: 10.1001/jamapsychiatry.2018.4156. PMID 30785624
- See also: Click here to visit the official website of the Body Dysmorphic Disorder Clinic at MGH — http://www.mghocd.org/bdd

RESULTS

PARTICIPANT FLOW:
Groups:
- Cognitive Behavior Therapy (CBT): Cognitive Behavior Therapy (CBT) is considered the psychosocial treatment of choice for BDD. It is a time-limited treatment that includes cognitive restructuring, mindfulness/attention retraining, exposure, and response prevention, specifically tailored for BDD. CBT is the only fully developed psychosocial treatment for BDD.
- Supportive Psychotherapy (SPT): SPT is a widely received psychosocial treatment by persons with BDD.
Period: Treatment Phase
Arm/Group | Cognitive Behavior Therapy (CBT) | Supportive Psychotherapy (SPT)
Started | 61 | 59
Completed | 44 | 48
Not Completed | 17 | 11
Not completed — Withdrawal by Subject | 13 | 10
Not completed — Suicidal Ideation | 2 | 0
Not completed — Need for higher level of care | 1 | 1
Not completed — Therapist conflict of interest | 1 | 0
Period: Follow-up
Arm/Group | Cognitive Behavior Therapy (CBT) | Supportive Psychotherapy (SPT)
Started | 44 | 48
Completed | 39 | 37
Not Completed | 5 | 11
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 5 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavior Therapy (CBT) | Supportive Psychotherapy (SPT) | Total
Number analyzed (Participants) | 61 | 59 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (14.5) | 33.4 (11.5) | 33.9 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 46 | 92
  Male | 15 | 13 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, Non-Hispanic | 47 | 53 | 100
  White, Hispanic | 2 | 2 | 4
  Black | 1 | 1 | 2
  Asian/Pacific Islander | 6 | 1 | 7
  Other | 5 | 2 | 7
Region of Enrollment [Count of Participants; unit: Participants] — Massachusetts General Hospital/Harvard Medical School and Rhode Island Hospital/Brown University will collaboratively recruited 120 adult participants to and were randomly assigned to receive CBT or SPT.
  Participants
    United States | 61 | 59 | 120

OUTCOME MEASURES:

1. Primary Outcome: Body Dysmorphic Disorder Symptoms (as Measured by the BDD-YBOCS)
Description: The Yale-Brown Obsessive Compulsive Scale Modified for BDD (BDD-YBOCS) is a 12-item, semi-structured, clinician-administered measure of BDD symptom severity. The scale's items are summed to yield a total score with a range from 0 to 48, with higher scores indicating more severe BDD symptoms. Treatment effects on BDD symptom severity were analyzed separately for the treatment period (i.e., weeks 0-24) and the follow-up period (i.e., weeks 24 to 50).
Time Frame: Change in BDD-YBOCS from baseline (week 0) to post-treatment (week 24), assessed every 4 weeks. Followup phase data was measured at week 37 and week 50.
Population: Intent to treat analysis on 120 subjects randomized to either CBT vs SPT. Some of the assessments visits were missed due to patient cancellations or study dropouts. The exact numbers analyzed are as specified below.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Cognitive Behavior Therapy (CBT): Cognitive-behavioral therapy (CBT) is a time-limited treatment that includes cognitive restructuring, mindfulness/attention retraining, exposure, and response prevention, specifically tailored for BDD.
- Supportive Psychotherapy (SPT): SPT is the most common psychosocial treatment received by persons with BDD.
Arm/Group | Cognitive Behavior Therapy (CBT) | Supportive Psychotherapy (SPT)
Number analyzed (Participants) | 61 | 59
score on a scale
  Baseline | 32.21 (4.72) | 31.49 (4.94)
  Week 4: number analyzed (Participants) | 52 | 55
  Week 4 | 26.92 (6.20) | 27.27 (6.41)
  Week 8: number analyzed (Participants) | 47 | 51
  Week 8 | 24.34 (7.70) | 25.09 (7.57)
  Week 12: number analyzed (Participants) | 43 | 46
  Week 12 | 19.67 (8.21) | 22.80 (8.90)
  week 16: number analyzed (Participants) | 42 | 46
  week 16 | 17.74 (9.21) | 22.13 (9.33)
  Week 20: number analyzed (Participants) | 44 | 43
  Week 20 | 15.95 (9.32) | 19.02 (9.44)
  Week 24: number analyzed (Participants) | 44 | 48
  Week 24 | 13.34 (9.46) | 18.67 (9.77)
  Week 37: number analyzed (Participants) | 43 | 41
  Week 37 | 12.30 (9.84) | 17.46 (9.81)
  Week 50: number analyzed (Participants) | 39 | 37
  Week 50 | 12.31 (10.75) | 16.90 (10.94)
Statistical Analysis 1: Comparison: Cognitive Behavior Therapy (CBT) vs Supportive Psychotherapy (SPT); We compared the difference in the rate of change in BDD symptom severity over time (during treatment phase) between the randomized treatment groups (CBT vs. SPT) using a latent growth curve model that included terms for treatment group, time, site, and all their interactions, modeling intercepts and slopes as random effects per person. Null hypothesis: The rate of change in BDD symptom severity in the CBT group will not be significantly different from the SPT group [to be tested]; Test type: Superiority; p < .01, Mixed Models Analysis — Degrees of freedom=90.9; Effect of interest: time by group interaction; Slope = -0.4602, Standard Error of Mean 0.1249 — The estimated value describes the mean slope difference of CBT compared to SPT
Statistical Analysis 2: Comparison: Cognitive Behavior Therapy (CBT) vs Supportive Psychotherapy (SPT); We compared the difference in the rate of change in BDD symptom severity over time (during the follow-up phase) between the randomized treatment groups (CBT vs. SPT) using a latent growth curve model that included terms for treatment group, time, site, and all their interactions, modeling intercepts and slopes as random effects per person. Null hypothesis: The rate of change in BDD symptom severity during follow-up will not differ significantly between CBT and SPT treatments [to be tested]; Test type: Superiority; p = .62, Mixed Models Analysis — Degrees of freedom=74.7; The effect of interest was the time by group interaction; Slope = -0.00984, Standard Error of Mean 0.1038 — The estimated value describes the mean slope difference of CBT compared to SPT during follow-up (week 24 to week 50)

2. Secondary Outcome: Insight Regarding BDD Beliefs (as Measured by the BABS)
Description: The Brown Assessment of Beliefs Scale (BABS) is a 7-item, semi-structured, clinician-administered measure that was used to assess insight regarding BDD-related beliefs (e.g., "I look deformed"). The first six items of the BABS were summed to obtain a total score ranging from 0 to 24, with higher scores reflecting poorer insight. Treatment effects on BABS score were analyzed separately for the treatment period (i.e., weeks 0-24) and the follow-up period (i.e., weeks 24 to 50).
Time Frame: Measured every 4 weeks during treatment, and at the 3-(wk 37) and 6-month(wk 50) follow-up visits
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavior Therapy (CBT) | Supportive Psychotherapy (SPT)
Number analyzed (Participants) | 61 | 59
units on a scale
  Baseline | 17.2459016 (4.2608909) | 15.4067797 (4.1817281)
  Week 4: number analyzed (Participants) | 52 | 55
  Week 4 | 14.7500000 (5.2538501) | 13.3090909 (5.0584463)
  Week 8: number analyzed (Participants) | 39 | 40
  Week 8 | 14.5128205 (5.9066056) | 12.8500000 (5.0765928)
  Week 12: number analyzed (Participants) | 43 | 46
  Week 12 | 10.8837209 (5.8562515) | 11.1304348 (6.0428422)
  week 16: number analyzed (Participants) | 42 | 46
  week 16 | 10.8571429 (7.2769983) | 9.7608696 (5.3465868)
  Week 20: number analyzed (Participants) | 39 | 36
  Week 20 | 9.8461538 (6.5435322) | 10.0277778 (5.8235292)
  Week 24: number analyzed (Participants) | 44 | 48
  Week 24 | 8.3636364 (7.5823875) | 7.9791667 (5.8908136)
  Week 37: number analyzed (Participants) | 43 | 41
  Week 37 | 6.6279070 (7.0000791) | 8.3170732 (5.8199614)
  Week 50: number analyzed (Participants) | 38 | 37
  Week 50 | 7.1578947 (7.9679300) | 7.3783784 (5.7848046)
Statistical Analysis 1: Comparison: Cognitive Behavior Therapy (CBT) vs Supportive Psychotherapy (SPT); We compared the change in Patient Insight over time (During Treatment phase) by randomized treatment group (CBT vs. SPT) using a latent growth curve model that included terms for treatment group, time, site, and all their interactions, modeling intercepts and slopes as random effects per person. Null hypothesis: The rate of improvement in insight in the CBT group will not be significantly different from the SPT group [to be tested]; Test type: Superiority; p = .10, Mixed Models Analysis — Degrees of freedom=93.2
Statistical Analysis 2: Comparison: Cognitive Behavior Therapy (CBT) vs Supportive Psychotherapy (SPT); We compared the change in Patient Insight over time (during the follow-up phase), by randomized treatment group (CBT vs. SPT) using a latent growth curve model that included terms for treatment group, time, site, and all their interactions, modeling intercepts and slopes as random effects per person. Null hypothesis: The rate of improvement in insight in the CBT group will not be significantly different from the SPT group during follow-up [to be tested]; Test type: Superiority; p = .45, Mixed Models Analysis — Degrees of freedom=74.5

3. Secondary Outcome: Depressive Symptoms (as Measured by the BDI-II)
Description: The Beck Depression Inventory-Second Edition (BDI-II) is a widely used 21-item self-report scale that assesses the severity of depressive symptoms during the past 2 weeks. Total scale scores range from 0 to 63, with higher scores indicating greater symptom severity. Treatment effects on depression were analyzed separately for the treatment period (i.e., weeks 0-24) and the follow-up period (i.e., weeks 24 to 50).
Time Frame: Measured every week during treatment, but analysis was performed only on BDI-II assessments close to assessment visits; wk 0, 4, 8, 12, 16, 20 and 24. Followup phase data was measured at week 37 and week 50.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavior Therapy (CBT) | Supportive Psychotherapy (SPT)
Number analyzed (Participants) | 61 | 59
units on a scale
  Baseline: number analyzed (Participants) | 61 | 58
  Baseline | 22.1639344 (13.1923972) | 22.8620690 (13.6117187)
  Week 4: number analyzed (Participants) | 52 | 57
  Week 4 | 18.6923077 (11.7215044) | 21.4035088 (14.9938793)
  Week 8: number analyzed (Participants) | 49 | 52
  Week 8 | 16.9591837 (13.4953066) | 19.3076923 (14.3178737)
  Week 12: number analyzed (Participants) | 45 | 48
  Week 12 | 15.2000000 (13.1037815) | 19.6041667 (14.8563900)
  week 16: number analyzed (Participants) | 45 | 48
  week 16 | 13.4000000 (12.9446374) | 17.5416667 (15.3220163)
  Week 20: number analyzed (Participants) | 44 | 43
  Week 20 | 11.4545455 (11.3474811) | 15.9302326 (14.2300744)
  Week 24: number analyzed (Participants) | 43 | 48
  Week 24 | 10.5348837 (12.2966291) | 15.6041667 (14.2541365)
  Week 37: number analyzed (Participants) | 39 | 36
  Week 37 | 9.2307692 (11.4120470) | 12.8611111 (13.9328036)
  Week 50: number analyzed (Participants) | 33 | 30
  Week 50 | 12.0606061 (15.3030622) | 13.6666667 (13.6541855)
Statistical Analysis 1: Comparison: Cognitive Behavior Therapy (CBT) vs Supportive Psychotherapy (SPT); We compared the change in depressive symptoms over time (During Treatment phase) by randomized treatment group (CBT vs. SPT) using a latent growth curve model that included terms for treatment group, time, site, and all their interactions, modeling intercepts and slopes as random effects per person. Null hypothesis: The rate of improvement in depressive symptoms in the CBT group will not be significantly different from the SPT group [to be tested]; Test type: Superiority; p = .05, Mixed Models Analysis — Degrees of freedom=89.1
Statistical Analysis 2: Comparison: Cognitive Behavior Therapy (CBT) vs Supportive Psychotherapy (SPT); We compared the change in depressive symptoms over time (during the follow-up phase), by randomized treatment group (CBT vs. SPT) using a latent growth curve model that included terms for treatment group, time, site, and all their interactions, modeling intercepts and slopes as random effects per person. Null hypothesis: The rate of change in depressive symptoms in the CBT group will not be significantly different from the SPT group during follow-up [to be tested]; Test type: Superiority; p = .26, Mixed Models Analysis — Degrees of freedom=63.7

4. Secondary Outcome: Life Satisfaction (Q-LESQ-SF)
Description: The Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form (Q-LESQ-SF) is a 16-item, self-report questionnaire that assesses life satisfaction over the past week. Questions 1-14 are then summed to a total score, and the total score is reported as a percentage maximum possible, such that the % score range is 0% to 100%, with higher scores indicating greater quality of life. Treatment effects on life satisfaction were analyzed separately for the treatment period (i.e., weeks 0-24) and the follow-up period (i.e., weeks 24 to 50).
Time Frame: Measured at week 0, 4, 12, 16, and 24 during treatment. Follow-up phase data was measured at week 37 and at week 50.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavior Therapy (CBT) | Supportive Psychotherapy (SPT)
Number analyzed (Participants) | 61 | 59
units on a scale
  Baseline: number analyzed (Participants) | 60 | 59
  Baseline | 48.7500000 (15.0603393) | 50.6961259 (16.6428814)
  Week 4: number analyzed (Participants) | 50 | 52
  Week 4 | 49.6648352 (15.8763522) | 51.7857143 (18.0729259)
  Week 12: number analyzed (Participants) | 42 | 45
  Week 12 | 61.0119048 (17.3217504) | 57.6190476 (17.6382690)
  Week 16: number analyzed (Participants) | 40 | 44
  Week 16 | 60.8894231 (15.9117634) | 57.3457792 (19.9192124)
  week 24: number analyzed (Participants) | 41 | 47
  week 24 | 68.2055749 (19.3905036) | 63.9437690 (19.0175684)
  Week 37: number analyzed (Participants) | 39 | 37
  Week 37 | 69.1849817 (17.5141781) | 64.3339768 (17.0683239)
  Week 50: number analyzed (Participants) | 36 | 30
  Week 50 | 66.5095899 (21.2768017) | 65.8928571 (19.3884669)
Statistical Analysis 1: Comparison: Cognitive Behavior Therapy (CBT) vs Supportive Psychotherapy (SPT); We compared the change in Quality of life satisfaction over time (During treatment phase) by randomized treatment group (CBT vs. SPT) using a latent growth curve model that included terms for treatment group, time, site, and all their interactions, modeling intercepts and slopes as random effects per person. Null hypothesis: The rate of change in Quality of life satisfaction severity in the CBT group will not be significantly different from the SPT group [to be tested]; Test type: Superiority; p = .04, Mixed Models Analysis — Degrees of freedom=91.4
Statistical Analysis 2: Comparison: Cognitive Behavior Therapy (CBT) vs Supportive Psychotherapy (SPT); We compared the change in the quality of life satisfaction over time (during the follow-up phase), by randomized treatment group (CBT vs. SPT) using a latent growth curve model that included terms for treatment group, time, site, and all their interactions, modeling intercepts and slopes as random effects per person. Null hypothesis: The rate of change in the quality of life satisfaction in the CBT group will not be significantly different from the SPT group during follow-up [to be tested]; Test type: Superiority; p = .82, Mixed Models Analysis — Degrees of freedom=74.7

5. Secondary Outcome: Treatment Credibility (Credibility/Expectancy Rating Scale)
Description: The Treatment Credibility/Expectancy Rating scale is a 4-item self-report questionnaire that assesses patients' judgments about the credibility of the treatment rationale, expectancy of change, and treatment acceptability. Treatment credibility is based on the mean score of the first three items, which are measured on 10-point Likert scales, so that mean scores range from 1 (lowest/worst) to 10 (highest/most). Treatment credibility was assessed at the baseline assessment (before treatment assignment) and after 1 month of treatment when patients are more familiar with the treatment protocol and rationale.
Time Frame: Measured twice during the study (week 0 [pre-treatment] and at week 4)
Population: The analysis population for this analysis was limited to those participants who completed the questionnaire (n=6 missing responses in the CBT arm, n=5 missing responses in the SPT arm at baseline), and decrease by week 4 due to study drop-out or missed assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Behavior Therapy (CBT) | Supportive Psychotherapy (SPT)
Number analyzed (Participants) | 55 | 54
score on a scale
  Week 0 | 7.10 (1.79) | 6.64 (1.84)
  Week 4: number analyzed (Participants) | 50 | 52
  Week 4 | 7.19 (1.68) | 6.28 (1.84)
Statistical Analysis 1: Comparison: Cognitive Behavior Therapy (CBT) vs Supportive Psychotherapy (SPT); Null hypothesis: There is no significant different in the perceived credibility of CBT and SPT; Test type: Superiority; p = 0.0095, ANOVA — Effect of interest: Treatment main effect, two-sided alpha = 0.05 effect adjusted for site effects, time effects, and interactions; repeated measures 3-way ANOVA (treatment type, site, time (repeated)) Effect of interest: main effect of treatment: F(num df=1, den df=112) = 5.17; Mean Difference (Net) = 0.7937, Standard Error of Mean 0.3007 — Least Squares Means difference

6. Secondary Outcome: Beliefs About Appearance (as Measured by the ASI-R)
Time Frame: Measured three times during the study (week 0 [pre-treatment], week 12, and week 24 [post-treatment])
Reporting Status: Not Posted

7. Secondary Outcome: Neuropsychological Functioning (as Measured by the ROCF)
Time Frame: Measured three times during the study (week 0 [pre-treatment], week 12, and week 24 [post-treatment])
Reporting Status: Not Posted

8. Secondary Outcome: Information Processing (as Measured by the ERT)
Time Frame: Measured three times during the study (week 0 [pre-treatment], week 12, and week 24 [post-treatment])
Reporting Status: Not Posted

9. Secondary Outcome: Sheehan Disability Scale (SDS)
Description: The Sheehan Disability Scale (SDS) is a 5-item self-report measure of functional impairment/disability. Items 1-3 (disability in work, social life/leisure, and family life/home responsibilities, respectively) are scored on Likert-scales that range from 0 (not at all) to 10 (extreme). The three items are then summed to yield an SDS total score, ranging from 0 (unimpaired) to 30 (highly impaired). Treatment effects on functional impairment were analyzed separately for the treatment period (i.e., weeks 0-24) and the follow-up period (i.e., weeks 24 to 50).
Time Frame: Measured at baseline, week 4, week 12, week 16, and week 24. Follow-up phase data was measured at week 37 and at week 50.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Behavior Therapy (CBT) | Supportive Psychotherapy (SPT)
Number analyzed (Participants) | 61 | 59
score on a scale
  Baseline: number analyzed (Participants) | 60 | 59
  Baseline | 16.3333333 (5.5621806) | 17.4406780 (6.0522757)
  Week 4: number analyzed (Participants) | 50 | 52
  Week 4 | 15.1000000 (6.3927574) | 15.5000000 (7.0056000)
  Week 12: number analyzed (Participants) | 42 | 45
  Week 12 | 11.7142857 (7.4023257) | 12.2222222 (7.8534558)
  Week 16: number analyzed (Participants) | 40 | 44
  Week 16 | 9.7250000 (7.6660674) | 11.7272727 (8.2019953)
  week 24: number analyzed (Participants) | 41 | 46
  week 24 | 7.9024390 (8.2970021) | 9.0869565 (7.2105666)
  Week 37: number analyzed (Participants) | 39 | 37
  Week 37 | 6.4871795 (6.3613628) | 9.2162162 (7.7428646)
  Week 50: number analyzed (Participants) | 36 | 30
  Week 50 | 6.6388889 (8.1980931) | 8.3666667 (7.8013409)
Statistical Analysis 1: Comparison: Cognitive Behavior Therapy (CBT) vs Supportive Psychotherapy (SPT); We compared the change in social functioning over time (During Treatment phase) by randomized treatment group (CBT vs. SPT) using a latent growth curve model that included terms for treatment group, time, site, and all their interactions, modeling intercepts, and slopes as random effects per person. Null hypothesis: The rate of improvement in social functioning in the CBT group will not be significantly different from the SPT group [to be tested]; Test type: Superiority; p = .30, Mixed Models Analysis — Degrees of freedom=88.0
Statistical Analysis 2: Comparison: Cognitive Behavior Therapy (CBT) vs Supportive Psychotherapy (SPT); We compared the change in social functioning over time (during the follow-up phase), by randomized treatment group (CBT vs. SPT) using a latent growth curve model that included terms for treatment group, time, site, and all their interactions, modeling intercepts and slopes as random effects per person. Null hypothesis: The rate of improvement in social functioning CBT group will not be significantly different from the SPT group during follow-up [to be tested]; Test type: Superiority; p = .85, Mixed Models Analysis — Degrees of freedom=74.5

10. Secondary Outcome: Treatment Satisfaction (CSQ-8)
Description: The Client Satisfaction Questionnaire (CSQ-8) is an 8-item self-report questionnaire that assesses satisfaction with clinical services received and has a score range of 8-32, where higher scores indicate higher satisfaction.
Time Frame: The CSQ-8 was assessed twice: at week 12 [mid-treatment] and at week 24 [post-treatment]
Population: The analysis population for this outcome was limited to those who were still in the study by week 12 (mid-treatmtent) and who completed the questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Behavior Therapy (CBT) | Supportive Psychotherapy (SPT)
Number analyzed (Participants) | 47 | 52
score on a scale
  Week 12: number analyzed (Participants) | 44 | 45
  Week 12 | 28.02 (2.88) | 26.60 (3.82)
  Week 24: number analyzed (Participants) | 42 | 48
  Week 24 | 29.40 (3.56) | 27.56 (4.07)
Statistical Analysis 1: Comparison: Cognitive Behavior Therapy (CBT) vs Supportive Psychotherapy (SPT); Null hypothesis: There is no significant difference in treatment satisfaction between patients with BDD assigned to CBT vs. SPT; Test type: Superiority; p = 0.0235, ANOVA — a priori significance level: 2-sided alpha = 0.05 effect adjusted for site effects, time effects, and interactions; repeated measures 3-way ANOVA (treatment type, site, time (repeated)) Effect of interest: main effect of treatment - F(num def=1,den df=79.9) = 15.55; Mean Difference (Net) = 1.5867, Standard Error of Mean 0.6882 — Least Squares Means difference

11. Secondary Outcome: Treatment Expectancy (Credibility/Expectancy Rating Scale)
Description: The Treatment Credibility/Expectancy Rating scale is a 4-item self-report questionnaire that assesses patients' judgments about the credibility of the treatment rationale, expectancy of change, and treatment acceptability. Treatment expectancy is a single item rating of "By the end of therapy, how much improvement in your anxiety do you think will occur?", rated on a scale from 0% to 100%. It was assessed at the baseline assessment (before treatment assignment) and after 1 month of treatment when patients are more familiar with the treatment protocol and rationale.
Time Frame: Measured twice during the study (week 0 [pre-treatment] and at week 4)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percent improvement expected (0-100%)
Arm/Group | Cognitive Behavior Therapy (CBT) | Supportive Psychotherapy (SPT)
Number analyzed (Participants) | 55 | 54
Percent improvement expected (0-100%)
  Week 0 | 58.36 (20.71) | 50.19 (19.28)
  Week 4: number analyzed (Participants) | 50 | 52
  Week 4 | 56.00 (20.40) | 46.73 (20.55)
Statistical Analysis 1: Comparison: Cognitive Behavior Therapy (CBT) vs Supportive Psychotherapy (SPT); Null hypotheses: There is no significant difference in patient expectancy of improvement between BDD patients assigned to CBT vs. SPT; Test type: Superiority; p = 0.0069, ANOVA — a priori significance level: 2-sided alpha=0.05 effect adjusted for site effects, time effects, and interactions; repeated measures 3-way ANOVA (treatment group, site, time (repeated)) effect of interest: main effect of treatment: F(num df=1, den df=110) = 7.59; Median Difference (Net) = 9.4390, Standard Error of Mean 3.4259 — Least Squares Mean difference

ADVERSE EVENTS:
Time Frame: Adverse event data was collected every 4 weeks at the beginning of therapy sessions, at the post-treatment visit, and at the 3- and 6-month follow-up visits (for a total of 1 year for each participant who completed the full study protocol). At these assessments, participants were probed for adverse events that occurred since the last adverse event assessment (usually 4 weeks prior).
Description: Participants were asked 4 questions about: (1) any major physical health problems or major physical injuries; (2) seeing a physical health or mental health provider for any reason; (3) any hospitalizations; or (4) any other major problems or concerns, all pertaining to the time since they were assessed last. Any "yes" resulted in a full event report. All serious adverse events are reported. Of non-serious events, only those affecting >5% in either treatment group are reported.
Arm/Group | Cognitive Behavior Therapy (CBT) | Supportive Psychotherapy (SPT)
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/59
Serious Adverse Events (participants affected / at risk) | 5/61 | 3/59
Other Adverse Events (participants affected / at risk) | 34/61 | 30/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Behavior Therapy (CBT) (N=61) | Supportive Psychotherapy (SPT) (N=59)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 1 (1)
Increase in BDD and depressive Symptoms (Psychiatric disorders) | 1 (2) | 0 (0) — Increase in BDD and depressive symptoms and relationship stressors.
Self-harm (Psychiatric disorders) | 1 (1) | 0 (0) — The participant cut himself/herself with a box cutter when distressed; was hospitalized.
Negative reaction to anesthesia (Gastrointestinal disorders) | 1 (1) | 0 (0) — The participant was hospitalized after a negative reaction to anesthesia. Symptoms included nausea and vomiting. The participant had received anesthesia for a more invasive procedure to address complications from a preexisting cyst.
Pain felt in one arm for a couple of days (General disorders) | 1 (1) | 0 (0) — The participant was admitted to an emergency room due to pain felt in one arm for a couple of days and was kept overnight for monitoring and released the next day with no official diagnosis given.
Mononucleosis (Infections and infestations) | 0 (0) | 1 (1) — Participant was hospitalized for one night for Mononucleosis (Mono) and was sick for 4 days.
Cardiac surgery (Cardiac disorders) | 1 (1) | 0 (0) — Cardiac surgery and recovery.
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1) — Anaphylactic shock
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Behavior Therapy (CBT) (N=61) | Supportive Psychotherapy (SPT) (N=59)
Increased anxiety and/or depression (Psychiatric disorders) | 8 (12) | 13 (14) — Increased depression or anxiety since starting study; no suicidal ideation.
Increase in other psychiatric symptoms (Psychiatric disorders) | 8 (8) | 3 (3) — Patients reported isolated occurrences of or temporary increases in other psychiatric symptoms, including obsessive thoughts, BDD symptoms, stress, fatigue, irritability, or binge drinking.
Suicidal ideation and/or self-harm (Psychiatric disorders) | 4 (6) | 1 (1) — Occurrences of suicidal ideation or incidents of self-harm (e.g., cutting)
Injury, poisoning, and procedural complications (Injury, poisoning and procedural complications) | 9 (16) | 5 (6) — AE descriptions included car accidents with minor injuries, broken or fractured bones, concussions, back injuries, accidental cut, ankle sprains, abrasion, alcohol poisoning, shoulder injury, cracked/chipped teeth, food poisoning, heat exhaustion
Nervous system disorders (Nervous system disorders) | 4 (4) | 3 (3) — AE descriptions included (flare up of) herniated disks, headaches, migraines, spine troubles, pinched nerve, and sharp pain in head.
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) — AE descriptions included flu, concerns about possible lung cancer (not detected), bronchitis, sore throat, and head and chest congestion.
Social circumstances (Social circumstances) | 2 (2) | 3 (3) — AE descriptions included friend dying in car crash, family conflict, spouse laid off from work, death of a parent, and hospitalization of a close family member.
Surgical and medical procedures (Surgical and medical procedures) | 2 (2) | 4 (4) — AE descriptions included minor outpatient surgery to to remove a splinter, cataract surgery, colonoscopy & ultrasound for removal of precancerous cells, scheduled surgeries, and a visit to a chiropractor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No